CLINICAL TRIAL: NCT01198080
Title: Bone Marrow Derived CD133+ Stem Cells Transplantation in Femoral Head Osteonecrosis
Brief Title: Evaluate the Effect of Bone Marrow Derived Cd133+ Cells in Patient With Osteonecrosis of Femoral Head
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-003
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2009-04

CONDITIONS: Osteonecrosis
Keywords: Avascular osteonecrosis,CD133+,core decompression
MeSH Terms: conditions — Osteonecrosis | interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- femoral osteonecrosis patients (Experimental): patientswith femoral head osteonecrosis
  Interventions: Biological: CD133+ cells

INTERVENTIONS:
Biological: CD133+ cells — bone marrow derived CD133+ cells injection with core compression
  Other Names: cell injection

SUMMARY:
Avascular necrosis is a disease where there is cellular death (necrosis) of bone components due to interruption of the blood supply. Without blood, the bone tissue dies and the bone collapses. If avascular necrosis involves the bones of a joint, it often leads to destruction of the joint articular surfaces. Avascular necrosis is especially common in the hip joint. A variety of methods are now used to treat avascular necrosis the most common being the total hip replacement, or THR.A new, more promising treatment is hip resurfacing or metal on metal (MOM) resurfacing.Another treatment is utilization of bone marrow derived stem cells.these stem cells can provide angiogenic factors and osteogenic cytokine to improve angiogenesis and bone formation.

DETAILED DESCRIPTION:
A vascular necrosis of femoral head is a debilitating disease resulting from interruption of blood supply to the bone. This pathologic process results in the death of marrow and osteocytes and, in its final stage, femoral head collapse. The most widespread treatment in the early stage of this disease is core decompression. This surgical procedure involves drilling into the femoral neck through the necrotic area, which reduces pressure within the bone and allows more blood vessels to form. This study is designed to evaluate the clinical safety and efficacy of CD133+ enriched bone marrow infusion adjacent with core decompression in patients with a vascular necrosis of femoral head . Patients will undergo core decompression followed by CD133+cell infusion into the cored area. Clinical assessment includes a MRI, Harries Hip Score,SF36, Visual Analogue Scale(VAS), and the WOMAC osteoarthritis Index.

ELIGIBILITY:
Inclusion Criteria:

* Upenn (Steinberg) classification of osteonecrosis, inclusive of Stages IIB and IIC. Diagnosis will be based on magnetic resonance imaging (MRI).
* Modified index of necrotic extent < 40
* Idiopathic and non-idiopathic osteonecrosis.
* No infection in affected bones at the time of surgery.
* Patient competent to give informed consent.
* Normal organ and marrow function defined as:

  * Leukocytes ≥ 3000/µL;
  * Absolute neutrophil count ≥ 1500/µL;
  * Platelets ≥ 140,000/µL;
  * Serum AST (SGOT)/ALT (SGPT) < 2.5 X institutional standard range;
  * Serum creatinine within normal limits, based on clinical laboratory normal range.
* Female patients not pregnant or lactating.
* Patients with a history of corticosteroids or on active therapy, will only be eligible for enrollment if corticosteroid use is suspended for 1 month prior and 6 months after cell therapy and surgery.
* Patients who have been treated with oral bisphosphonates are eligible for the trial if treatment was stopped at least 6 months prior to enrollment.

Exclusion Criteria:

* Stages IA, IB, IC, IIA, IIIA or more severe femoral head osteonecrosis, primarily based on diagnosis by MRI.
* Flattening of the femur head (UPenn Stage IV) or articular cartilage collapse at the time of core decompression surgery.
* Septic arthritis; stress fracture, or non-osteonecrosis metabolic bone diseases (e.g., Paget's disease of bone, osteogenesis imperfecta, primary hyperparathyroidism, fibrous dysplasia [monostotic, polyostotic McCune-Albright syndrome] and osteopetrosis).
* Any active bisphosphonate treatment or any history of intravenous (IV) treatment
* HIV, syphilis, positive at time of screening.
* Active hepatitis B or hepatitis C infection at the time of screening
* Known allergies to protein products (horse or bovine serum, or porcine trypsin).
* Patients who will require continuous, systemic, high dose corticosteroid therapy (more than 7.5 mg/day) within 6 months after surgery.
* received chemotherapy, radiotherapy or immunotherapy in the past 2 years.
* Immunodeficiency diseases.
* Participation in another clinical study in the past 30 days or concurrent participation in another clinical trial.
* History of regular alcohol consumption exceeding 2 drinks/day (1 drink = 5 oz [150 mL] of wine or 12 oz [360 mL] of beer or 1.5 oz [45 mL] of hard liquor) within 6 months of screening and/or history of illicit drug use.
* MRI-incompatible internal devices (pacemakers, aneurysm clips, etc)
* Body mass index (BMI) of 40 Kg/m2 or greater
* Patients unable to tolerate general anesthesia defined as an American Society of Anesthesiologists (ASA) criteria of > 2
* Patients with poorly controlled diabetes mellitus (HbA1C > 8%), or with peripheral neuropathy, or known concomitant vascular problems.
* Patients receiving treatment with hematopoietic growth factors or anti-vasculogenesis or anti-angiogenesis treatment
* Traumatic osteonecrosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
safety of bone marrow derived CD133+ cells transplantation | 6 months
  Evaluation safety of bone marrow CD133+ cells transplantation in patients with osteonecrosis of femoral head

SECONDARY OUTCOMES:
improve patient quality of life | 12 months
  evaluate the ability of bone marrow derived CD133+ cells to improve patient quality of life
decrease hip articular change | 24 month
  evaluate the ability of bone marrow derived CD133+ cells to decrease hip articular change
side effects | 24 months
  Evaluate side effects of bone marrow derived CD133+ cells transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Ahmad Vosough, MD, Principal Investigator — Board scientific; Nasser Aghdami, MD,PhD, Principal Investigator — Head of regenerative medicine center; Mohammad Reza Baghban Eslami, PhD, Study Director — Board Sientific; mohssen Emadeddin, MD, Principal Investigator — Orthopedic Investigator
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org